CLINICAL TRIAL: NCT05403372
Title: Evaluation of an Implant Free Interatrial Shunt to Improve Heart Failure
Acronym: EASE HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: InterShunt Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-004
Record Dates: First submitted 2022-05-24; First posted 2022-06-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- InterShunt PAS-C (Experimental)
  Interventions: Device: PAS-C System

INTERVENTIONS:
Device: PAS-C System — The InterShunt PAS-C System is a transcatheter system that creates a shunt by excising tissue from the interatrial septum resulting in a left to right atrial shunt that off-loads elevated left atrial pressure, potentially reducing symptoms and improving quality of life. The PAS-C System does not require a permanent implant to maintain patency of the interatrial shunt.

SUMMARY:
This is a prospective, single arm feasibility study to establish safety and performance of the PAS-C System in subjects with heart failure and elevated left atrial pressure.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented chronic, symptomatic heart failure and NYHA Class II, Class III or ambulatory Class IV at the time of screening visit and receiving guideline directed medical therapy.
* At least one hospitalization or emergency department visit with heart failure as the primary or secondary diagnosis or intravenous diuretic treatment for heart failure or documentation of elevated BNP.
* LVEF ≥ 40%.
* Echocardiographic evidence of diastolic dysfunction during the baseline echocardiography:
* Per baseline exercise right heart catheterization, site measured elevated left atrial pressure with a gradient compared to right atrial pressure.

Key Exclusion Criteria:

* Stroke or thromboembolic event in the past 6 months.
* Severe or advanced heart failure such as Stage D heart failure, non-ambulatory NYHA Class IV, cardiac index less than 2.0 L/min/m2, LVEDD > 6 cm, or received inotropic therapy for LVEF less than 40% within 6 months prior to enrollment.
* Any of the following within 3 months prior to enrollment: myocardial infarction, percutaneous cardiac intervention, CABG, cardiac resynchronization therapy, AICD, or indicated for coronary revascularization at the time of enrollment.
* More than moderate valve disease (mitral, tricuspid, aortic) at the time of enrollment.
* Chronic pulmonary disease requiring continuous home oxygen or hospitalization within prior 12 months for pulmonary disease.
* BMI > 40.
* 6-minute Walk Test distance less than 100 m or greater than 450 m performed during baseline screening, or unable to perform baseline bicycle exercise test.
* Any of the following at the time of baseline screening: moderate or worse right heart dysfunction, requires dialysis, atrial fibrillation with ventricular rate > 100 bpm, systolic blood pressure greater than 170 mmHg (average of 3 measurements at baseline).
* Evidence of precapillary pulmonary hypertension defined as PVR > 2 Wood units at rest, TPG > 15 at rest or with exercise, resting RA > 15 mmHg, or RA to PCWP ratio > 0.7 at rest and with exercise.
* Anatomic anomaly that precludes creation of interatrial shunt.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who experience a major adverse cardiac or cerebrovascular event (MACCE) or systemic embolization. | 1 month
  The proportion of subjects who experience a composite MACCE or systemic embolization event.

SECONDARY OUTCOMES:
Echocardiogram evidence of interatrial shunt with left to right atrial flow | 1 month
  Proportion of subjects with visible shunt demonstrating left to right atrial flow as determined by echocardiographer

CONTACTS AND LOCATIONS:
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No